CLINICAL TRIAL: NCT06140355
Title: cHAnging the Perceived Pain INtensity in divErSe Populations With Spinal Cord Injury
Brief Title: HAPPINESS: cHAnging the Perceived Pain INtEnSity in Populations With Spinal Cord Injury and With Health Disparities: A Feasibility Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: PT-2023-32452
Record Dates: First submitted 2023-11-07; First posted 2023-11-20 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries | interventions — Qigong

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): adults with SCI-related neuropathic pain with at least 50% from diverse groups randomized to experimental group
  Interventions: Behavioral: Qigong
- Active comparison group (Active Comparator): adults with SCI-related neuropathic pain with at least 50% from diverse groups randomized to active comparator group
  Interventions: Behavioral: Daily 2 min pain management survey

INTERVENTIONS:
Behavioral: Qigong — a Qigong introduction class and a 12-week remote Qigong intervention, with a 6-month follow-up
  Arms: Experimental group
Behavioral: Daily 2 min pain management survey — Completing one short survey (2 min) daily through your phone or computer (you will get a survey link through email or text), with a 6-month follow-up.
  Arms: Active comparison group

SUMMARY:
Chronic neuropathic pain affects 69% of adults with spinal cord injury (SCI). Current treatment options are limited (primarily pain medications) with insufficient benefits and significant risks for addiction and adverse effects. Of the available mind and body approaches, Qigong is the most accessible for adults with SCI with evidence for effectiveness in reducing pain, but there is insufficient evidence to make recommendations for adults with SCI. Thus, the feasibility of Qigong in SCI needs to be established.

To support our feasibility study, we investigated a 12-week remote Qigong program in adults with SCI and neuropathic pain. We recruited 23 adults with SCI, 18 completed the study, and 12 completed the 1-year follow-up. They practiced Qigong 138% of the required intensity (which was, at least 3x/week with Qigong video through the internet). Their pain was reduced by 44% after 12 weeks of Qigong practice and was still reduced at the 6-week and 1-year follow-up. However, three key elements need to be addressed before performing a larger effectiveness study: (1) feasibility/acceptability of Qigong from adults with SCI of diverse backgrounds; (2) feasibility of the study design with control group); and (3) objective outcome measures.

This R34 feasibility study, the HAPPINESS trial (cHAnging the Perceived Pain INtensity in divErSe populations with Spinal cord injury), will expand on our prior study to consolidate feasibility with a rigorous protocol. We will address the following aims: AIM 1. Identify the facilitators/barriers to participating in a Qigong study through focus groups/interviews with stakeholders from diverse backgrounds, defined as Hispanics, veterans, and adults living in rural, underserved areas. AIM 2. Establish the feasibility of study design/methods of the HAPPINESS trial in adults with SCI (at least 50% of diverse backgrounds) through pre-specified targets for recruitment/enrollment, feasibility, and acceptability of design and outcomes. Using a Phase I randomized controlled trial design, 40 adults with SCI-related neuropathic pain will be randomized to 12-week remote Qigong intervention OR a short daily pain management survey that can be completed on phone/iPad/computer + 6-month follow-up. The study results will facilitate a rigorous structure to design larger effectiveness studies and facilitate a clear pathway for researchers to investigate Qigong and other mind-body approaches for whole-person health in diverse groups of adults with chronic/neurological disorders.

ELIGIBILITY:
Inclusion Criteria:

* 18+ years old
* medically stable
* with neuropathic pain 4 or above on the numeric pain rating scale + screened with painDETECT
* willing to participate in a remote Qigong intervention (from any location with internet connection)
* fluent in English or Spanish
* access to the internet and a computer/iPad or smartphone

Exclusion Criteria:

* uncontrolled seizure disorder
* cognitive impairment and/or communicative disability (e.g., due to brain injury) preventing them from following directions or from learning
* ventilator dependency
* major medical complications
* pressure ulcers hindering prolonged sitting or lying down
* (planning to become) pregnant or planning a major surgery during the study (given study duration, regular Qigong practice, and frequent check-ins)
* regular Tai Chi or Qigong practice in the past 6 months (3x/week or more)
* currently engaged in other rehabilitation programs that would influence outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-08-20 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
recruitment rates | 6 months post-intervention
  The proportion of potential participants contacted who agreed to participate
the recruitment rate for complete and incomplete SCI | 6 months post-intervention
  Ratio of complete/incomplete SCI.
Attrition rates in Qigong and Manage My Pain app group. | 6 months post-intervention
  Proportion of people withdrawing from the study in either group. Drop-out due to unrelated reasons will count as part of the general attrition.
intervention adherence | 6 months post-intervention
  the website log times will indicate the date and duration that the video is accessed. From this information, we will collect the number of minutes that they practice.
  This information will be checked with the self-report during the weekly calls, in which they will report the number of minutes per week they have practiced.
the frequency of use of the Manage My Pain app (recommended daily check in) | 6 months post-intervention
  Weekly/ monthly check-ins (reporting min/week of practice) to identify facilitators and barriers to practicing Qigong. The website logs time and duration of video access. A Qigong certified instructor will do 1:1 Qigong session with each participant via zoom monthly for quality control/to give guidance.
Feasibility of adhering to the collection of quantitative measure 1 | 6 months post-intervention
  % Adherence in completing all assessments during the study and in the monthly follow-up phase
Feasibility of adhering to the collection of quantitative measure 2 | 6 months post-intervention
  % Adherence to wearing Fitbit Charge 6 and sending the data through their phone App

CONTACTS AND LOCATIONS:
Overall Officials: Ann Van de Winckel, PhD, MSPT, PT, Principal Investigator — University of Minnesota
Locations (3):
- United States (3):
  - University of Miami, Miami, Florida
  - University of Minnesota, Minneapolis, Minnesota
  - University of Texas - Rio Grande Valley, Harlingen, Texas

REFERENCES:
- [Derived] Van de Winckel A, Zhang L, Lim KO, Morse LR, Woodliff B, Maestre G, Baker K. Changing the Perceived Pain Intensity in Populations With Spinal Cord Injury and With Health Disparities (HAPPINESS): Protocol for a Feasibility Study. JMIR Res Protoc. 2025 Nov 19;14:e82431. doi: 10.2196/82431. PMID 41259096